CLINICAL TRIAL: NCT04357249
Title: Outcome of Capsular After Pediatric Cataract Surgery With Primary Intraocular Lens Implantation
Acronym: Capsular
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, yin ying zhao [yyzhao], Wenzhou Medical University
Other Study IDs: FYN-capsular
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pediatric Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the outcome of capsular in children with cataract, and to explore potential preoperative structural clues for postoperative glaucoma. The investigators included children with cataract planning to have cataract surgery in our institute. Exclusion criteria were: a history of ocular trauma, a history of intraocular surgery, preoperative glaucoma, steroid use before surgery, a history of maternal rubella syndrome, chronic anterior uveitis, persistent fetal vasculature, ocular anomalies associated with an increased risk of glaucoma, unable to complete examinations. The investigators recorded age at surgery, gender and relevant ocular and systemic histories. All patients underwent slit lamp biomicroscopy, slit lamp adapted anterior segment photography.All patients were examined at 1 week, 1 month, 3 months, 6 months, 1 year, 18 months, and two years after surgery. Patients were followed for two years or until the development of severe VAO requiring Nd: YAG laser capsulotomy, whichever came first. The examinations consisted of visual acuity, IOP measurement by a Tonopen tonometer (Reichert, Inc., Seefeld, Germany), fundoscopy, an assessment by high-resolution digital retroillumination imaging (detailed protocol presented below).The primary outcomes were the areas of the posterior capsular opening at different postoperative follow-up visits and during operation.A paired T test was used to compare the areas of the PCO between the postoperative visits and baseline.

ELIGIBILITY:
Inclusion Criteria:

Participants included eyes of children with unilateral or bilateral cataract.

Exclusion Criteria:

Patients with glaucoma, ocular trauma, corneal disorders, persistent hyperplastic primary vitreous, rubella, Lowe syndrome, capsular fibrosis, or surgical complications, as well as those whose pupils could not dilate normally postoperation or who could not complete the follow-up, were excluded.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants included eyes of children with unilateral or bilateral cataract.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-03-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
area of PCO | 2015.5.1- 2020.8-1
  area of posterior capsular opening

CONTACTS AND LOCATIONS:
Overall Officials: ZHAO YUNE, MD, Study Director — executive dean
Locations (1):
- Wenzhou Medical Colledge, Wenzhou, Zhejiang, China